CLINICAL TRIAL: NCT03851289
Title: Combination of Platelet-Rich Fibrin and Calcium Sulfate in Socket Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr CHEAH CHIA WEI, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DF RD 1621/0076 (L)
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Tooth Extraction
Keywords: socket augmentation; platelet-rich fibrin; calcium sulfate; xenograft
MeSH Terms: interventions — Calcium Sulfate; Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test (PRF-CS) (Experimental): After atraumatic tooth extraction, the socket was gently curettage and irrigated with saline. Combination of platelet-rich fibrin and calcium sulfate was placed into the socket followed by a PRF plug . Black silk suture (3-0) was placed on mesial, mid and distal using simple interrupted technique.
  Interventions: Combination Product: platelet-rich fibrin and calcium sulfate
- control (PRF-X) (Active Comparator): After atraumatic tooth extraction, the socket was gently curettage and irrigated with saline. Combination of platelet-rich fibrin and xenograft (MinerOss® X) was placed into the socket followed by a PRF plug . Black silk suture (3-0) was placed on mesial, mid and distal using simple interrupted technique.
  Interventions: Combination Product: platelet-rich fibrin and xenograft

INTERVENTIONS:
Combination Product: platelet-rich fibrin and calcium sulfate
  Arms: test (PRF-CS)
Combination Product: platelet-rich fibrin and xenograft
  Arms: control (PRF-X)

SUMMARY:
This study evaluated the effectiveness of socket grafting material, combination of plate-rich fibrin and calcium sulfate. 5 subjects were grafted with this material, 5 subjects were grafted with combination of plate-rich fibrin and xenograft.

DETAILED DESCRIPTION:
Calcium sulfate (CS), an alloplastic material, is widely accepted as a socket grafting material and undergoes rapid and complete resorption. Studies have shown that CS creates an osteoconductive lattice that stimulates bone ingrowth into a defect. PRF poses multiple growth factors, anti-inflammatory cytokines and adhesion molecules. It is biologically active up to one week. The combination of these 2 materials will serve as good grafting material for tooth socket, in order to preserve vertical and horizontal dimensions.

ELIGIBILITY:
Inclusion Criteria:

* maxillary premolar teeth requiring extraction
* neighboring mesial and distal sound/restored teeth present
* alveolar bone level (measured from periapical radiographs) more than 50% of the root length
* age ranges from 25-55 years

Exclusion Criteria:

* bony fenestration of the socket wall confirmed from CBCT scan
* acute signs of infection
* periodontally compromised teeth
* absence of buccal plates
* any systemic disease which may hinder the healing process

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
vertical dimension at baseline | before extraction
  measurements were done on radiograph (CBCT) images
horizontal dimension at baseline | before extraction
  measurements were done on radiograph (CBCT) images
soft tissue level at baseline | before extraction
  measurements were done on stone models
volume at baseline | before extraction
  measurements were done on radiograph (CBCT) images

SECONDARY OUTCOMES:
vertical dimension after extraction | five months after extraction
  measurements were done on radiograph (CBCT) images
horizontal dimension after extraction | five months after extraction
  measurements were done on radiograph (CBCT) images
soft tissue level after extraction | five months after extraction
  measurements were done on stone models
volume after extraction | five months after extraction
  measurements were done on radiograph (CBCT) images

CONTACTS AND LOCATIONS:
Overall Officials: CHIA W CHEAH, Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: No
socio demographic background

REFERENCES:
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Darby I, Chen ST, Buser D. Ridge preservation techniques for implant therapy. Int J Oral Maxillofac Implants. 2009;24 Suppl:260-71. PMID 19885449
- [Background] Cardaropoli D, Cardaropoli G. Preservation of the postextraction alveolar ridge: a clinical and histologic study. Int J Periodontics Restorative Dent. 2008 Oct;28(5):469-77. PMID 18990998
- [Background] Fickl S, Zuhr O, Wachtel H, Stappert CF, Stein JM, Hurzeler MB. Dimensional changes of the alveolar ridge contour after different socket preservation techniques. J Clin Periodontol. 2008 Oct;35(10):906-13. doi: 10.1111/j.1600-051X.2008.01305.x. Epub 2008 Aug 17. PMID 18713258
- [Background] Jambhekar S, Kernen F, Bidra AS. Clinical and histologic outcomes of socket grafting after flapless tooth extraction: a systematic review of randomized controlled clinical trials. J Prosthet Dent. 2015 May;113(5):371-82. doi: 10.1016/j.prosdent.2014.12.009. Epub 2015 Mar 4. PMID 25749077
- [Background] Anwandter A, Bohmann S, Nally M, Castro AB, Quirynen M, Pinto N. Dimensional changes of the post extraction alveolar ridge, preserved with Leukocyte- and Platelet Rich Fibrin: A clinical pilot study. J Dent. 2016 Sep;52:23-9. doi: 10.1016/j.jdent.2016.06.005. Epub 2016 Jun 20. PMID 27338946
- [Background] Guarnieri R, Pecora G, Fini M, Aldini NN, Giardino R, Orsini G, Piattelli A. Medical grade calcium sulfate hemihydrate in healing of human extraction sockets: clinical and histological observations at 3 months. J Periodontol. 2004 Jun;75(6):902-8. doi: 10.1902/jop.2004.75.6.902. PMID 15295959
- [Background] Strocchi R, Orsini G, Iezzi G, Scarano A, Rubini C, Pecora G, Piattelli A. Bone regeneration with calcium sulfate: evidence for increased angiogenesis in rabbits. J Oral Implantol. 2002;28(6):273-8. doi: 10.1563/1548-1336(2002)0282.3.CO;2. PMID 12498535
- [Background] Simon BI, Gupta P, Tajbakhsh S. Quantitative evaluation of extraction socket healing following the use of autologous platelet-rich fibrin matrix in humans. Int J Periodontics Restorative Dent. 2011 Jun;31(3):285-95. PMID 21556385
- [Background] Dohan Ehrenfest DM, de Peppo GM, Doglioli P, Sammartino G. Slow release of growth factors and thrombospondin-1 in Choukroun's platelet-rich fibrin (PRF): a gold standard to achieve for all surgical platelet concentrates technologies. Growth Factors. 2009 Feb;27(1):63-9. doi: 10.1080/08977190802636713. PMID 19089687
- [Background] Cheah CW, Vaithilingam RD, Siar CH, Swaminathan D, Hornbuckle GC. Histologic, histomorphometric, and cone-beam computerized tomography analyses of calcium sulfate and platelet-rich plasma in socket preservation: a pilot study. Implant Dent. 2014 Oct;23(5):593-601. doi: 10.1097/ID.0000000000000148. PMID 25192162
- [Background] Yilmaz S, Karaca EO, Ipci SD, Cakar G, Kuru BE, Kullu S, Horwitz J. Radiographic and histologic evaluation of platelet-rich plasma and bovine-derived xenograft combination in bilateral sinus augmentation procedure. Platelets. 2013;24(4):308-15. doi: 10.3109/09537104.2012.695033. Epub 2012 Jun 21. PMID 22720715
- [Background] Potres Z, Deshpande S, Kloeppel H, Voss K, Klineberg I. Assisted Wound Healing and Vertical Bone Regeneration with Simultaneous Implant Placement: A Histologic Pilot Study. Int J Oral Maxillofac Implants. 2016 Jan-Feb;31(1):45-54. doi: 10.11607/jomi.3951. PMID 26800162
- [Background] Manavella V, Romano F, Corano L, Bignardi C, Aimetti M. Three-Dimensional Volumetric Changes in Severely Resorbed Alveolar Sockets After Ridge Augmentation with Bovine-Derived Xenograft and Resorbable Barrier: A Preliminary Study on CBCT Imaging. Int J Oral Maxillofac Implants. 2018 March/April;33(2):373-382. doi: 10.11607/jomi.5684. Epub 2017 Aug 17. PMID 28817739
- [Background] Aimetti M, Manavella V, Corano L, Ercoli E, Bignardi C, Romano F. Three-dimensional analysis of bone remodeling following ridge augmentation of compromised extraction sockets in periodontitis patients: A randomized controlled study. Clin Oral Implants Res. 2018 Feb;29(2):202-214. doi: 10.1111/clr.13099. Epub 2017 Nov 17. PMID 29148597
- [Background] Pang C, Ding Y, Zhou H, Qin R, Hou R, Zhang G, Hu K. Alveolar ridge preservation with deproteinized bovine bone graft and collagen membrane and delayed implants. J Craniofac Surg. 2014 Sep;25(5):1698-702. doi: 10.1097/SCS.0000000000000887. PMID 25148644
- [Background] Das S, Jhingran R, Bains VK, Madan R, Srivastava R, Rizvi I. Socket preservation by beta-tri-calcium phosphate with collagen compared to platelet-rich fibrin: A clinico-radiographic study. Eur J Dent. 2016 Apr-Jun;10(2):264-276. doi: 10.4103/1305-7456.178298. PMID 27095909
- [Background] Zhang Y, Ruan Z, Shen M, Tan L, Huang W, Wang L, Huang Y. Clinical effect of platelet-rich fibrin on the preservation of the alveolar ridge following tooth extraction. Exp Ther Med. 2018 Mar;15(3):2277-2286. doi: 10.3892/etm.2018.5696. Epub 2018 Jan 4. PMID 29456635
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Background] Hauser F, Gaydarov N, Badoud I, Vazquez L, Bernard JP, Ammann P. Clinical and histological evaluation of postextraction platelet-rich fibrin socket filling: a prospective randomized controlled study. Implant Dent. 2013 Jun;22(3):295-303. doi: 10.1097/ID.0b013e3182906eb3. PMID 23644909
- [Background] Aimetti M, Romano F, Griga FB, Godio L. Clinical and histologic healing of human extraction sockets filled with calcium sulfate. Int J Oral Maxillofac Implants. 2009 Sep-Oct;24(5):902-9. PMID 19865631
- [Background] Kalash S, Aboelsaad N, Shokry M, Choukroun J. The efficiency of using advanced PRF-xenograft mixture around immediate implants in the esthetic zone: a randomized controlled clinical trial. Journal of Osseointegration. 9(4):317-22, 2017
- [Background] Barone A, Ricci M, Romanos GE, Tonelli P, Alfonsi F, Covani U. Buccal bone deficiency in fresh extraction sockets: a prospective single cohort study. Clin Oral Implants Res. 2015 Jul;26(7):823-30. doi: 10.1111/clr.12369. Epub 2014 Mar 31. PMID 24684275
- [Background] Intini G, Andreana S, Margarone JE 3rd, Bush PJ, Dziak R. Engineering a bioactive matrix by modifications of calcium sulfate. Tissue Eng. 2002 Dec;8(6):997-1008. doi: 10.1089/107632702320934092. PMID 12542945
- [Background] Calasans-Maia M, Resende R, Fernandes G, Calasans-Maia J, Alves AT, Granjeiro JM. A randomized controlled clinical trial to evaluate a new xenograft for alveolar socket preservation. Clin Oral Implants Res. 2014 Oct;25(10):1125-30. doi: 10.1111/clr.12237. Epub 2013 Aug 13. PMID 23937306
- [Background] Clark D, Rajendran Y, Paydar S, Ho S, Cox D, Ryder M, Dollard J, Kao RT. Advanced platelet-rich fibrin and freeze-dried bone allograft for ridge preservation: A randomized controlled clinical trial. J Periodontol. 2018 Apr;89(4):379-387. doi: 10.1002/JPER.17-0466. PMID 29683498
- [Background] Lekovic V, Kenney EB, Weinlaender M, Han T, Klokkevold P, Nedic M, Orsini M. A bone regenerative approach to alveolar ridge maintenance following tooth extraction. Report of 10 cases. J Periodontol. 1997 Jun;68(6):563-70. doi: 10.1902/jop.1997.68.6.563. PMID 9203100
- [Background] Cardaropoli G, Araujo M, Lindhe J. Dynamics of bone tissue formation in tooth extraction sites. An experimental study in dogs. J Clin Periodontol. 2003 Sep;30(9):809-18. doi: 10.1034/j.1600-051x.2003.00366.x. PMID 12956657
- [Background] Dohan Ehrenfest DM, Pinto NR, Pereda A, Jimenez P, Corso MD, Kang BS, Nally M, Lanata N, Wang HL, Quirynen M. The impact of the centrifuge characteristics and centrifugation protocols on the cells, growth factors, and fibrin architecture of a leukocyte- and platelet-rich fibrin (L-PRF) clot and membrane. Platelets. 2018 Mar;29(2):171-184. doi: 10.1080/09537104.2017.1293812. Epub 2017 Apr 24. PMID 28437133
- [Background] Clark RA. Fibrin and wound healing. Ann N Y Acad Sci. 2001;936:355-67. doi: 10.1111/j.1749-6632.2001.tb03522.x. PMID 11460492
- [Background] Dohan Ehrenfest DM, Rasmusson L, Albrektsson T. Classification of platelet concentrates: from pure platelet-rich plasma (P-PRP) to leucocyte- and platelet-rich fibrin (L-PRF). Trends Biotechnol. 2009 Mar;27(3):158-67. doi: 10.1016/j.tibtech.2008.11.009. Epub 2009 Jan 31. PMID 19187989
- [Background] Thakkar DJ, Deshpande NC, Dave DH, Narayankar SD. A comparative evaluation of extraction socket preservation with demineralized freeze-dried bone allograft alone and along with platelet-rich fibrin: A clinical and radiographic study. Contemp Clin Dent. 2016 Jul-Sep;7(3):371-6. doi: 10.4103/0976-237X.188567. PMID 27630503
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Amarnath GS, Kumar U, Hilal M, Muddugangadhar BC, Anshuraj K, Shruthi CS. Comparison of Cone Beam Computed Tomography, Orthopantomography with Direct Ridge Mapping for Pre-Surgical Planning to Place Implants in Cadaveric Mandibles: An Ex-Vivo Study. J Int Oral Health. 2015;7(Suppl 1):38-42. PMID 26225103
- [Background] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Vignoletti F, Matesanz P, Rodrigo D, Figuero E, Martin C, Sanz M. Surgical protocols for ridge preservation after tooth extraction. A systematic review. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:22-38. doi: 10.1111/j.1600-0501.2011.02331.x. PMID 22211304
- [Background] Ten Heggeler JM, Slot DE, Van der Weijden GA. Effect of socket preservation therapies following tooth extraction in non-molar regions in humans: a systematic review. Clin Oral Implants Res. 2011 Aug;22(8):779-88. doi: 10.1111/j.1600-0501.2010.02064.x. Epub 2010 Nov 22. PMID 21091540
- [Background] Avila-Ortiz G, Elangovan S, Kramer KW, Blanchette D, Dawson DV. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):950-8. doi: 10.1177/0022034514541127. Epub 2014 Jun 25. PMID 24966231
- [Background] Iocca O, Farcomeni A, Pardinas Lopez S, Talib HS. Alveolar ridge preservation after tooth extraction: a Bayesian Network meta-analysis of grafting materials efficacy on prevention of bone height and width reduction. J Clin Periodontol. 2017 Jan;44(1):104-114. doi: 10.1111/jcpe.12633. Epub 2016 Dec 5. PMID 27712001
- [Background] Tomasi C, Sanz M, Cecchinato D, Pjetursson B, Ferrus J, Lang NP, Lindhe J. Bone dimensional variations at implants placed in fresh extraction sockets: a multilevel multivariate analysis. Clin Oral Implants Res. 2010 Jan;21(1):30-6. doi: 10.1111/j.1600-0501.2009.01848.x. PMID 20070744
- [Background] Araujo M, Linder E, Lindhe J. Effect of a xenograft on early bone formation in extraction sockets: an experimental study in dog. Clin Oral Implants Res. 2009 Jan;20(1):1-6. doi: 10.1111/j.1600-0501.2008.01606.x. PMID 19126101
- [Background] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L, Cardaropoli G. Socket preservation using bovine bone mineral and collagen membrane: a randomized controlled clinical trial with histologic analysis. Int J Periodontics Restorative Dent. 2012 Aug;32(4):421-30. PMID 22577648
- [Background] Abraham S, Deepak K, Ambili R, Preeja C, Archana V. Gingival biotype and its clinical significance-A review. The Saudi Journal for Dental Research. 5(1):3-7, 2014
- [Background] Lee SA, Kim AC, Prusa LA Jr, Kao RT. Characterization of dental anatomy and gingival biotype in Asian populations. J Calif Dent Assoc. 2013 Jan;41(1):31-3, 36-9. PMID 23437604
- [Background] Fernandez RF, Bucchi C, Navarro P, Beltran V, Borie E. Bone grafts utilized in dentistry: an analysis of patients' preferences. BMC Med Ethics. 2015 Oct 20;16(1):71. doi: 10.1186/s12910-015-0044-6. PMID 26486125
- [Derived] Sultan T, Cheah CW, Ibrahim NB, Asif MK, Vaithilingam RD. Three-dimensional assessment of the extraction sockets, augmented with platelet-rich fibrin and calcium sulfate: A clinical pilot study. J Dent. 2020 Oct;101:103455. doi: 10.1016/j.jdent.2020.103455. Epub 2020 Aug 21. PMID 32828845

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT03851289/Prot_SAP_001.pdf